CLINICAL TRIAL: NCT00335582
Title: The EPIC (Evaluating Perioperative Ischemia Reduction by Clonidine) Study: A Randomized, Double-blinded Trial of Clonidine for Reducing Cardiac Morbidity and Mortality Following Non-cardiac Surgery.
Brief Title: EPIC (Evaluating Perioperative Ischemia Reduction by Clonidine)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Anesthesiologists' Society (Other)
Responsible Party: Dr. Duminda Wijeysundera, Toronto General Hospital, University Health Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REB#05-0146-B
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-05

CONDITIONS: Heart Disease
Keywords: alpha 2 agonists; cardiac events; non cardiac surgery
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: clonidine hydrochloride — One hour prior to surgery, patients randomized to the treatment arm will receive clonidine as both a 0.2 mg oral tablet and 0.2 mg/day transdermal patch patch will be removed on postoperative day 4 (or hospital discharge, whichever is earlier)

SUMMARY:
In Canada 1 patient in 200 dies within 30 days of an operation. More than half of these deaths are the direct result of a heart related complication. This cause of death happens 4 times more often than in the same people who do not have an operation. We do not have an effective way to stop these heart attacks. Stress causes the heart rate and the blood pressure to go up which causes the heart to work harder and may be the reason for some heart attacks. One group of drugs that stops the heart from working harder and decrease the number of heart related complications are BETA-BLOCKERS. We wish to add another drug, which has been shown to reduce heart rate and blood pressure, will reduce the number of heart attacks after an operation. CLONIDINE has been shown to reduce heart attacks after operations. Since we know it is not a good idea to stop beta-blockers we want to see if giving clonidine as well as a beta-blocker is safe and has the desired effect of decreasing the number of heart attacks. We want to find out how good the combination of these two drugs are at decreasing the number of heart attacks.

Hypothesis: The addition of clonidine to chronic b-blockade will reduce mortality and cardiac morbidity among intermediate-to-high risk patients undergoing non-cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 45 years
2. Current use of b-blocker therapy>=30 days prior to surgery
3. Undergoing non-cardiac surgery with an expected length of stay ≥ 48 hours for medical reasons
4. Informed consent
5. Undergoing major vascular surgery (excluding carotid endarterectomy, dialysis shunt, and vein stripping) OR

Meet >= 2of the following criteria:

1. Coronary artery disease
2. Congestive heart failure
3. Stroke or transient ischemic attack
4. Diabetes mellitus requiring oral hypoglycemic or insulin therapy
5. Preoperative renal insufficiency (creatinine clearance below 60 mL/min)
6. Peripheral vascular disease, as defined by any of the following: history of ischemic intermittent claudication or rest pain, history of revascularization procedure to legs, peripheral arterial obstruction of >= 50% luminal diameter
7. Age >=70 years
8. Intermediate-risk surgical procedure: intra-peritoneal, intra-thoracic, carotid endarterectomy, major orthopedic (hip, knee, spine) surgery, radical prostatectomy, or head-and-neck surgery

Exclusion criteria: - if meets any of the following

1. Prior adverse reaction to clonidine or a-2 agonists
2. Current use of Clonidine or a-2 agonists
3. Current congestive heart failure
4. Only b-blocker taken by patient is sotalol
5. Left ventricular ejection fraction <=40%
6. Systolic blood pressure < = 90 mmHg
7. Concomitant life-threatening disease likely to limit life expectancy to <=30 days.
8. Clinically significant aortic stenosis, defined as an aortic valve area <=1.0 cm2 and/or peak trans-valvular pressure gradient >= 25 mmHg

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2006-06; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
To preform feasibility study looking at the safety and efficacy of adding clonidine to chronic b-blockade on patient-relevant outcomes (mortality, myocardial infarction, prolonged hospitalization) in large randomized controlled trials | Daily until discharge and 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Duminda Wijeysundera, MD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Wijeysundera DN, Choi PT, Badner NH, Brasher PM, Dresser GK, Delgado DH, Beattie WS. A randomized feasibility trial of clonidine to reduce perioperative cardiac risk in patients on chronic beta-blockade: the EPIC study. Can J Anaesth. 2014 Nov;61(11):995-1003. doi: 10.1007/s12630-014-0226-6. Epub 2014 Sep 5. PMID 25189430